CLINICAL TRIAL: NCT00540579
Title: A Phase I/II Study of CC-4047 in Combination With Gemcitabine in Subjects With Untreated Advanced Carcinoma of the Pancreas
Brief Title: CC-4047 With Gemcitabine for Untreated Advanced Carcinoma of the Pancreas
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: SCRI Development Innovations, LLC (Other)
Collaborators: Celgene Corporation (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SCRI GI 105; PO-PANC-PI-009
Record Dates: First submitted 2007-10-05; First posted 2007-10-08 (Estimated); Results first posted 2013-03-13 (Estimated); Last update posted 2013-03-13 (Estimated); Status verified 2013-02

CONDITIONS: Pancreatic Cancer
Keywords: Pancreas; Untreated; Advanced; Gemcitabine; CC-4047
MeSH Terms: conditions — Pancreatic Neoplasms | interventions — pomalidomide; Gemcitabine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Intervention (Experimental): All patients received gemcitabine 1000 mg/m2 IV on days 1, 8, and 15 of a 28 day cycle. Pomalidomide was administered orally on days 1-21 at doses escalated from 2 mg to 10 mg daily.
  Interventions: Drug: Pomalidomide; Drug: Gemcitabine

INTERVENTIONS:
Drug: Pomalidomide — Phase 1: Subjects will be enrolled in dose-escalating cohorts to be treated with CC-4047 on days 1-21 Phase II: Subjects will be enrolled to receive oral CC-4047 at the MTD days 1 - 21
  Other Names: CC-4047
Drug: Gemcitabine — 1000 mg/m2 IV on days 1, 8, and 15 of 28 day cycle
  Other Names: Gemzar

SUMMARY:
Because the activity of CC-4047 addresses numerous mechanisms of carcinoma growth inhibition - including, but not limited to anti-angiogenesis - CC-4047 has been selected for development as part of induction chemotherapy regimens for solid tumors. This study in pancreatic cancer is designed to determine the appropriate CC-4047 dose and regimen in combination with gemcitabine.

DETAILED DESCRIPTION:
Phase I

Primary:

• To determine the maximum tolerated dose (MTD) and evaluate the safety profile of oral CC-4047 given on days 1-21 in combination with gemcitabine on days 1, 8, and 15 every 28 days in subjects with advanced pancreatic carcinoma.

Secondary:

• To explore the anti-tumor activity of the combination of CC-4047 and gemcitabine as combination therapy in subjects with advanced pancreatic carcinoma.

Phase II

Primary:

• To explore the anti-tumor activity of the combination of CC-4047 on days 1-21 and gemcitabine on days 1, 8, and 15 every 28 days in subjects with advanced pancreatic carcinoma.

Secondary:

• To evaluate the safety profile of the combination of CC-4047 and gemcitabine as combination therapy in subjects with advanced pancreatic carcinoma.

ELIGIBILITY:
Inclusion Criteria:

1. Understand and voluntarily sign an informed consent form.
2. Age ≥ 18 years at the time of signing the informed consent form.
3. Must be able to adhere to the study visit schedule and other protocol requirements.
4. Histological or cytological documentation of adenocarcinoma of the pancreas with metastases not amenable to curative surgery or definitive radiation. Patients with locally advanced disease are not eligible.
5. Radiographic or clinical evidence of measurable advanced metastatic pancreatic carcinoma. Subjects must have measurable disease according to the international criteria proposed by the Response Evaluation Criteria in Solid Tumors (RECIST) Committee for target lesions (see Appendix 14.2).
6. Subjects may have been previously treated with adjuvant radiation therapy and 5-fluorouracil or Gemzar as a radiosensitizer in the adjuvant setting if they currently have evidence of progression. Following completion of XRT, no further adjuvant chemotherapy with either Gemzar or 5-FU is permitted. No prior Gemzar® for metastatic disease or for primary treatment of locally advanced disease is allowed. Gemzar® used solely as a radiation sensitizer in the adjuvant setting is permitted.
7. ECOG performance status of 0 or 1.
8. Females of childbearing potential (FCBP)† must have a negative serum or urine pregnancy test with a sensitivity of at least 50 mIU/mL 10 - 14 days prior to and again within 24 hours of starting CC-4047 and must either commit to continued abstinence from heterosexual intercourse or begin TWO acceptable methods of birth control, one highly effective method and one additional effective method AT THE SAME TIME, at least 4 weeks before she starts taking CC-4047. FCBP must also agree to ongoing pregnancy testing. Men must agree not to father a child and agree to use a condom if his partner is of child bearing potential. All patients must be counseled at a minimum of every 28 days about pregnancy precautions and risks of fetal exposure (see Appendix 14.6).

Exclusion Criteria:

1. Pregnant or lactating females.
2. Any serious medical condition or psychiatric illness that prevents the study subject from signing the informed consent form or places the study subject at an unacceptable risk if he or she participates in the study.
3. Prior therapy with CC-4047, lenalidomide, or thalidomide.
4. Prior use of systemic therapy for the treatment of adenocarcinoma of the pancreas with the exception of 5-fluorouracil or Gemzar® as a radiosensitizer in the adjuvant setting
5. Concurrent use of any other anti-cancer agents.
6. Any of the following laboratory abnormalities:

   * Absolute neutrophil count (ANC) < 1,500 cells/mm3 (1.5 x 109/L)
   * Platelet count < 100,000 cells/ mm3 (100 x 109/L)
   * Serum creatinine > 2.5 mg/dL (221 μmol/L)
   * Serum SGOT/AST or SGPT/ALT > 3.0 x upper limit of normal (ULN); in case of liver metastases > 5 x ULN
   * Serum total bilirubin > 2.0 mg/dL (34 μmol/L)
7. Surgery or radiation therapy within 14 days of study enrollment as outlined below.

   * Surgery within 14 days of the start of study (patients must have recovered from effects of surgery; 7 days may be considered for minor procedures).
   * Palliative radiation therapy within 14 days of the start of study. The radiation therapy may not be to the only site of measurable disease. Adjuvant therapy is permitted in accordance with the inclusion criteria.
8. Prior history of malignancy (except basal cell or squamous cell carcinoma or carcinoma in situ of the cervix or breast, localized prostate cancer with PSA < 1.0 mg/dL) unless the subject has been free of disease for ≥ 3 years.
9. Known brain or leptomeningeal disease (CT scan or MRI of the brain required only in case of clinical suspicion of central nervous system involvement).
10. Grade ≥ 2 neuropathy.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 23 (Actual)
Dates: Start 2007-11; Primary Completion 2008-12 (Actual); Study Completion 2011-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jeffrey Infante, M.D., Study Chair — SCRI Development Innovations, LLC
Locations (2):
- United States (2):
  - University of Colorado Cancer Center, Aurora, Colorado
  - Tennessee Oncology, PLLC, Nashville, Tennessee

REFERENCES:
- [Background] Infante JR, Jones SF, Bendell JC, Spigel DR, Yardley DA, Weekes CD, Messersmith WA, Hainsworth JD, Burris HA 3rd. A phase I, dose-escalation study of pomalidomide (CC-4047) in combination with gemcitabine in metastatic pancreas cancer. Eur J Cancer. 2011 Jan;47(2):199-205. doi: 10.1016/j.ejca.2010.09.002. Epub 2010 Nov 2. PMID 21051221

RESULTS

PARTICIPANT FLOW:
Groups:
- Pomalidomide/Gemcitabine: All patients received gemcitabine 1000 mg/m2 IV on days 1, 8, and 15 of a 28 day cycle. Pomalidomide was administered orally on days 1-21 at doses escalated from 2 mg to 10 mg daily.
Period: Overall Study
Arm/Group | Pomalidomide/Gemcitabine
Started | 23
Completed | 23
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Pomalidomide/Gemcitabine
Number analyzed (Participants) | 23
Age Continuous [Median (Full Range); unit: years] | 62 [47 to 78]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 7
  Male | 16
Region of Enrollment [Number; unit: participants]
  United States | 23

OUTCOME MEASURES:

1. Primary Outcome: Determination of Maximum Tolerated Dose (MTD), The Dose of Study Drug(s) Which Causes <33% of Patients Treated to Experience Unacceptable Side Effects
Description: Unacceptable side effects or dose-limiting toxicities (DLTs) were defined as follows:
  * Inability to Complete cycle 1 of therapy due to drug-related toxicity.
  * > Grade 3 non-hematological drug-related toxicity (excluding alopecia) despite optimal supportive care
  * Febrile neutropenia (absolute neutrophil count [ANC] <1,000/μL and fever >101° F (38.5° C))
  * Grade 4 neutropenia that occurs prior to day 21. (Grade 4 neutropenia that occurs after day 21 but resolves within 7 days of the scheduled cycle 2, will not be considered DLT)
  * Platelet count < 25,000/μL
  * Inability to initiate Cycle 2, Day 1 therapy within 7 days of scheduled start (i.e. cannot delay the start of Cycle 2 by more than 7 days following the normal 7 day recovery period) due to drug-related toxicity.
Time Frame: 6 months
Population: Two patients withdrew consent and were unevaluable for DLT. One patient suffered subdural hematoma (non-treatment related) and was unevaluable for DLT.
Measure: Number; unit: milligrams
Arm/Group | Pomalidomide/Gemcitabine
Number analyzed (Participants) | 20
milligrams
  Pomalidomide | 10
  Gemcitabine | 1000

2. Primary Outcome: The Safety and Tolerability of Protocol Treatment, Defined as the Percentage of Patients Experiencing Severe or Life-threatening Side Effects Per CTCAE Version 3.0
Description: The relative incidence of Grade 3/4 adverse events from protocol treatment as defined by Common Terminology Criteria for Adverse Events v3.0 (CTCAE)
Time Frame: 24 Months
Population: All patients treated with pomalidomide and gemcitabine were assessed for Grade 3/4 toxicities
Measure: Number (95% Confidence Interval); unit: percentage of patients
Arm/Group | Pomalidomide/Gemcitabine
Number analyzed (Participants) | 23
percentage of patients | 39 [19.07 to 58.93]

ADVERSE EVENTS:
Arm/Group | Pomalidomide/Gemcitabine
Serious Adverse Events (participants affected / at risk) | 13/23
Other Adverse Events (participants affected / at risk) | 23/23
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Pomalidomide/Gemcitabine (N=23)
Constipation (Gastrointestinal disorders) | 1 (1)
Hyperglycemia (Metabolism and nutrition disorders) | 1 (1)
ARDS (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Perforation, GI (Gastrointestinal disorders) | 1 (1)
GI - Other (Gastrointestinal disorders) | 1 (1) — Gastroparesis
Obstruction - GI (Gastrointestinal disorders) | 1 (1)
Hematoma (Blood and lymphatic system disorders) | 1 (1)
Hemorrhage - GI (Gastrointestinal disorders) | 1 (1)
Febrile Neutropenia (General disorders) | 1 (1)
Pain (General disorders) | 1 (1)
Infection - Pneumonia (Infections and infestations) | 1 (1)
Thrombosis/Thrombus/Embolism (Vascular disorders) | 4 (4)
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Renal - Other (Renal and urinary disorders) | 1 (1) — Pyelonephritis
Infection - Skin (Infections and infestations) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Pomalidomide/Gemcitabine (N=23)
Abdominal Pain (General disorders) | 6 (7)
ALT (Metabolism and nutrition disorders) | 2 (5)
Hemoglobin (Blood and lymphatic system disorders) | 12 (45)
Anorexia (Gastrointestinal disorders) | 7 (7)
Arthralgia (Musculoskeletal and connective tissue disorders) | 2 (3)
Ascites (Gastrointestinal disorders) | 4 (5)
AST (Metabolism and nutrition disorders) | 3 (4)
Atrial Fibrillation (Cardiac disorders) | 2 (2)
Back Pain (General disorders) | 6 (6)
Alkaline Phosphatase (Metabolism and nutrition disorders) | 3 (3)
Bone Pain (General disorders) | 2 (3)
Chills (General disorders) | 4 (5)
Constipation (Gastrointestinal disorders) | 10 (11)
Cough (Respiratory, thoracic and mediastinal disorders) | 4 (4)
Dehydration (Gastrointestinal disorders) | 4 (5)
Diarrhea (Gastrointestinal disorders) | 9 (18)
Dizziness (Nervous system disorders) | 5 (6)
Dry Mouth (Gastrointestinal disorders) | 2 (2)
Dysgeusia (Gastrointestinal disorders) | 2 (2)
Dyspepsia (Gastrointestinal disorders) | 2 (2)
Fatigue (General disorders) | 14 (20)
Flatulence (Gastrointestinal disorders) | 4 (4)
Hyperuricemia (gout) (Metabolism and nutrition disorders) | 2 (2)
Headache (General disorders) | 3 (3)
Hyperglycemia (Metabolism and nutrition disorders) | 2 (2)
Sweating (General disorders) | 3 (3)
Hypokalemia (Metabolism and nutrition disorders) | 3 (5)
Hypotension (Cardiac disorders) | 3 (3)
Nausea (Gastrointestinal disorders) | 8 (11)
Peripheral Neuropathy (Nervous system disorders) | 2 (2)
Neutrophils (Blood and lymphatic system disorders) | 12 (81)
Night Sweats (General disorders) | 2 (2)
Peripheral Edema (Blood and lymphatic system disorders) | 10 (15)
Pain - Extremity (General disorders) | 3 (3)
Polyuria (Renal and urinary disorders) | 2 (2)
Pruritis (Skin and subcutaneous tissue disorders) | 2 (2)
Thrombus/Thrombosis/Embolism (Vascular disorders) | 8 (10)
Fever (General disorders) | 6 (12)
Rash (Skin and subcutaneous tissue disorders) | 11 (16)
Nasal/Paranasal Reaction (Respiratory, thoracic and mediastinal disorders) | 2 (3)
Syncope (Nervous system disorders) | 2 (2)
Platelets (Blood and lymphatic system disorders) | 9 (20)
Blurred Vision (Eye disorders) | 2 (2)
Vomiting (Gastrointestinal disorders) | 7 (11)
Weight Loss (Gastrointestinal disorders) | 2 (2)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The sponsor can review/embargo results communications prior to public release for a period that is >60 days but ≤180 days from date submitted to sponsor, who may require changes to the communication in order to remove specifically identified confidential information (other than study data) and/or delay the proposed publication to enable the sponsor to seek patent protection for inventions. The PI may not publish its results until 18 mos. after the trial has been completed at all sites.